CLINICAL TRIAL: NCT02657252
Title: Polidocanol Versus Glucose For Sclerotherapy Treatment Of Telangiectasia Of The Lower Limbs: Protocol For A Randomized, Controlled Clinical Trial
Brief Title: Polidocanol Versus Glucose Treatment of Telangiectasia Trial
Acronym: PG3T
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Dr Matheus Bertanha, Assistant professor, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPECLIN
Record Dates: First submitted 2016-01-07; First posted 2016-01-15 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-11

CONDITIONS: Varicose Veins; Telangiectasis
Keywords: telangiectasis; varicose veins; veins; glucose; sclerotherapy
MeSH Terms: conditions — Varicose Veins; Telangiectasis | interventions — Glucose; Polidocanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucose (Active Comparator): An application session 0.2% Polidocanol + 70% Glucose to treat telangiectasis of the lower limb selected, with a maximum volume of 5 ml. Return to a week to investigate the adverse effects and 2 months for proof of efficacy and adverse effects
  Interventions: Drug: Glucose
- Polidocanol with Glucose (Active Comparator): An application session 0.2% Polidocanol + 70% Glucose to treat telangiectasis of the lower limb selected, with a maximum volume of 5 ml. Return to a week to investigate the adverse effects and 2 months for proof of efficacy and adverse effects
  Interventions: Drug: Polidocanol with Glucose

INTERVENTIONS:
Drug: Glucose — Sclerotherapy of telangiectasis in one lower limb.
  Other Names: Hypertonic dextrose
  Arms: Glucose
Drug: Polidocanol with Glucose — Sclerotherapy of telangiectasis in one lower limb.
  Other Names: Asclera; Varithena
  Arms: Polidocanol with Glucose

SUMMARY:
It will be done a randomized triple-blind study comparing 0,2% polidocanol versus 75% hypertonic glucose of sclerotherapy in lower limbs´ telangiectasis. It will be included only adult women with reticular veins on the side of the thighs and mild venous insufficiency (CEAP 1). The primary endpoint will be efficacy, and secondary will be safety.

DETAILED DESCRIPTION:
Background. The prevalence of chronic venous disease is high in the general population, mainly in young women, and in milder cases the usual complaint is aesthetic. Various techniques are used for treatment of mild varicose disease, including surgical treatment, laser ablation and sclerotherapy. Telangiectasis are those with less than 1 mm diameter, reddish and important contribution to the aesthetic damage, and sometimes they are related to local pain. There is no consensus in the literature about the effectiveness of treatment with sclerotherapy, despite of being an usual procedure with different chemicals.

Methods and design. One hundred lower limbs of healthy women between 18 and 65 years will be triple blind randomized to receive treatment with polidocanol 0.2% diluted in 70% hypertonic glucose versus 75% hypertonic glucose for sclerotherapy treatment of telangiectasis. The patients will be examined and clinically classified. It will be included patients with telangiectasis sited at out's thigh, and only one extremity will be included per patient. The patients with varicose disease CEAP 2 or more will not be included. The treatment will be carried out in only one session and the medication volume not exceeding 5 ml. Clinical follow-up protocols will be filled on regular visits on days 0 - 7 - 60 concomitantly with photograph documentation. Supplementary examination for venous mapping with ultrasound pretreatment is performed for all patients.

Discussion. This prospective controlled double-blind randomized trial aims to verify and compare the efficacy and safety for sclerotherapy treatment of telangiectasis of the lower limbs. The results may help physicians to choose the best sclerotherapy treatment for telangiectasis.

ELIGIBILITY:
Inclusion Criteria:

* females
* with telangiectasis on thigh side
* clinical classification of chronic venous disease C1(mild venous disease),
* minimum age of 18 year-old and maximum age 65 year-old
* agreement with the study
* signing the free and informed consent ( IC)
* not use anticoagulant drugs .

Exclusion Criteria:

* male
* varicose disease in any quantity or location with clinical classification of chronic venous disease different of C1(mild venous disease)
* restrict mobility
* arterial insufficiency
* be allergic to any substance that may be related to the study drugs
* any cause of dermatitis on application site
* don´t be free of comorbidities clinically serious as diabetes mellitus, heart failure, respiratory failure, uncontrolled hypertension with medication, and uncontrolled hypothyroidism
* pregnancy
* previous deep vein thrombosis (DVT)
* family history of DVT
* thrombophilia
* do not agree with the search terms

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matheus Bertanha, Dr, Principal Investigator — Botucatu School of Medicine
Locations (1):
- Vascular Lab, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bertanha M, Camargo PA, Moura R, Yoshida WB, Pimenta RE, Mariuba JV, Alcantara GP, de Paula DR, Sobreira ML. Polidocanol versus glucose in the treatment of telangiectasia of the lower limbs (PG3T): Protocol for a randomized, controlled clinical trial. Medicine (Baltimore). 2016 Sep;95(39):e4812. doi: 10.1097/MD.0000000000004812. PMID 27684809

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some patients (n=17) were withdrawn because did not appear at the previous scheduled appointments, and were replaced for new ones. In order to avoid loss of individuals we have decided to include 17 more patients.
Units Other Than Participants: lower limbs
Period: Overall Study
Arm/Group | Glucose | Polidocanol With Glucose
Started | 57; 57 lower limbs | 58; 58 lower limbs
Completed | 47; 47 lower limbs | 51; 51 lower limbs
Not Completed | 10; 10 lower limbs | 7; 7 lower limbs

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glucose | Polidocanol With Glucose | Total
Number analyzed (Participants) | 57 | 58 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 58 | 115
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (10) | 43.6 (10) | 42.2 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 115
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — The patients were from Botucatu (or nearby), São Paulo, Brazil
  Participants
    Brazil | 57 | 58 | 115

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Extent of Telangiectasias
Description: Efficiency in promoting the disappearance of the treated telangiectasias, making the comparison between the initial measurements in centimeters and after two months, then comparing the treatment between the two treatments
Time Frame: 2 months
Population: Only one lower limb submited to the treatment.
Measure: Mean (Standard Deviation); unit: percent of change negative values
Arm/Group | Glucose | Polidocanol With Glucose
Number analyzed (Participants) | 47 | 51
percent of change negative values | 57.24 (22.69) | 76.08 (18.63)

2. Secondary Outcome: Skin Hyperpigmentation
Description: Observed after two months of treatment the occurrence of hyperpigmentation stains in the treated areas. Measuring in centimeters those stains and compare the two treatments together.
Time Frame: 2 months
Measure: Median (95% Confidence Interval); unit: percentage of hyperpigmentation
Arm/Group | Glucose | Polidocanol With Glucose
Number analyzed (Participants) | 47 | 51
percentage of hyperpigmentation | 0.49 [0 to 13.15] | 0 [0 to 10.85]

3. Secondary Outcome: Number of Participants With Deep Venous Thrombosis (DVT)
Description: Observe after one week of treatment occurred if clinical signs and symptoms of deep vein thrombosis (DVT) and perform duplex ultrasound for confirmation. Compare the results between the two groups to establish a security policy.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Glucose | Polidocanol With Glucose
Number analyzed (Participants) | 47 | 51
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Right after two months post procedure
Description: Hyperpigmentation: Linear measure above the projection area of hyperpigmentation post procedure. The length of this line was provided by the Image J software (ImageJ is a public domain, Java-based image processing program developed at the National Institutes of Health)
Arm/Group | Glucose | Polidocanol With Glucose
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/51
Other Adverse Events (participants affected / at risk) | 28/47 | 21/51
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glucose (N=47) | Polidocanol With Glucose (N=51)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 28 | 21 — Hyperpigmentation is a pigmented line that can occurred after sclerotherapy treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes